CLINICAL TRIAL: NCT06902792
Title: A Single-Center, Single-Arm, Phase I Clinical Trial of Adebrelimab Combined With Trametinib in the Treatment of Refractory Recurrent Langerhans Cell Histiocytosis in Children and Adolescents
Brief Title: Adebrelimab Combined With Trametinib in the Treatment of Refractory Recurrent Langerhans Cell Histiocytosis in Children and Adolescents
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2025-06-103
Record Dates: First submitted 2025-03-10; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Histiocytosis, Langerhans-Cell
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab (Experimental): Phase 1, 1 case in total
  Subject 1:
  This study marks the first application of Adebrelimab in pediatric patients with Langerhans Cell Histiocytosis (LCH). The initial dose is 20 mg/kg, delivered via a 60-minute intravenous infusion. If no Dose-Limiting Toxicity (DLT) occurs, the second dose of 20 mg/kg will be administered in the second cycle. Treatment cycles consist of dosing every 4 weeks, up to a maximum of 6 cycles.
  Phase 2, 2-5 cases in total
  Subjects 2 and 3:
  If the first subject exhibits no DLT, the second and third subjects will be enrolled and receive 20 mg/kg of Adebrelimab on day 1. Treatment cycles will last 4 weeks, with dosing administered every 4 weeks, for up to 6 cycles.
  Subjects 4-6:
  If one DLT occurs among the first three subjects, three additional subjects will be enrolled and given 20 mg/kg of Adebrelimab. If two or more DLTs occur among the first three subjects, three additional subjects will be enrolled and administered a reduced dose of 10 mg/kg.
  Interventions: Drug: treated group

INTERVENTIONS:
Drug: treated group — This study marks the first application of Adebrelimab in pediatric patients with Langerhans Cell Histiocytosis (LCH). The initial dose is 20 mg/kg, delivered via a 60-minute intravenous infusion. If no Dose-Limiting Toxicity (DLT) occurs, the second dose of 20 mg/kg will be administered in the second cycle. Treatment cycles consist of dosing every 4 weeks, up to a maximum of 6 cycles.

SUMMARY:
Phase 1, 1 case in total

Subject 1:

This study marks the first application of Adebrelimab in pediatric patients with Langerhans Cell Histiocytosis (LCH). The initial dose is 20 mg/kg, delivered via a 60-minute intravenous infusion. If no Dose-Limiting Toxicity (DLT) occurs, the second dose of 20 mg/kg will be administered in the second cycle. Treatment cycles consist of dosing every 4 weeks, up to a maximum of 6 cycles.

Phase 2, 2-5 cases in total

Subjects 2 and 3:

If the first subject exhibits no DLT, the second and third subjects will be enrolled and receive 20 mg/kg of Adebrelimab on day 1. Treatment cycles will last 4 weeks, with dosing administered every 4 weeks, for up to 6 cycles.

Subjects 4-6:

If one DLT occurs among the first three subjects, three additional subjects will be enrolled and given 20 mg/kg of Adebrelimab. If two or more DLTs occur among the first three subjects, three additional subjects will be enrolled and administered a reduced dose of 10 mg/kg.

Following the successful completion of these phases, a subsequent phase will commence to further assess the efficacy and safety of Adebrelimab and fulfill the biological research objectives.

DETAILED DESCRIPTION:
1. Research and treatment period 1) Pre-treatment: Patients receive trametinib for 1-2 weeks (maximum 2 weeks) based on tumor load. For those with a poor treatment response (defined as at least one Disease Activity Score, excluding blood markers, greater than 1), cytarabine (100mg/m² once daily) is administered via 12-hour continuous infusion for 2-4 days, starting on day 11.

2) Combination therapy: Each cycle lasts 28 days. Adebrelimab is administered on day 1, and trametinib is given on days 22-28. This regimen is repeated for 6 cycles.

3) Medication regimen and dosage adjustment:

1. Trametinib dosing: For patients < 6 years, the dose is 0.032 mg/kg/day; for patients ≥ 6 years, the dose is 0.025 mg/kg/day. It is administered on days 1-7. No dose adjustments are required, but treatment should be permanently discontinued in cases of Grade 4 complications, including but not limited to deep vein thromboembolism, pulmonary embolism, an absolute decrease in LVEF >20% from baseline, or retinal vein occlusion.
2. Adebrelimab dosing: The dose is 20 mg/kg per administration, titrated over 60 minutes.

   2. Availability of investigational drugs/treatments
   1. Trametinib is manufactured by GlaxoSmithKline Manufacturing S.p.A.. Company address: VIA A.FLEMING, 2-VERONA 37135.ITALIA (Italy). Imported drug registration number: H20190068, H20190069.
   2. Adebrelimab is manufactured by Suzhou Shengdia Bio-pharmaceutical Co., Ltd, No. 350 Fengli Street, Suzhou Industrial Park, Suzhou Area, Pilot Free Trade Zone, China (Jiangsu), State Drug License No. S20233106.

      -Generic Name: Adebrelimab Injection

      -Trade name: Ariel

      -English name: Adebrelimab Injection

      -Hanyu Pinyin: Adebeili Dankang Zhusheye

      -Active ingredient: Adebrelimab is a humanized monoclonal antibody targeting programmed death ligand 1 (PD-L1).

      -Excipients:Sucrose, Succinic Acid, Sodium Hydroxide, Polysorbate 80 and Water for Injection.
      * Properties:The product is a clear liquid, ranging from colorless to light yellow.
      * Specifications: 600 mg(12ml)/vial

        3.ministration Method and Dosage Adjustment

   <!-- -->

   1. Method of administration The infusion should be administered over 30 to 60 minutes, with a maximum infusion time of 2 hours. Intravenous administration is contraindicated for this product.
   2. Drug Configuration

      Dilution and Preparation Instructions:

      This product is intended for intravenous administration and must be diluted and dispensed by a healthcare professional:

      -Visually inspect Adebrelimab Injection for particulate matter or discoloration prior to use. The solution should appear colorless to pale yellow. Do not use if particulate matter or discoloration is observed.

      -Withdraw the required dose from Adebrelimab Injection and slowly inject it into an infusion bag containing 0.9% Sodium Chloride Injection or 5% Glucose Injection. Gently invert the bag to ensure thorough mixing. The final diluted concentration should range from 0.5 mg/mL to 9 mg/mL. As this product lacks preservatives, aseptic techniques must be strictly followed during preparation.

      -This product is for single use only. Discard any unused portion of the vial.
      * Dispose of unused medication or waste materials in compliance with local regulations.
   3. Infusion rate The infusion should be administered over 30 to 60 minutes, with a maximum infusion duration of 2 hours. Intravenous administration is contraindicated for this product.
   4. Precautions for Infusion An infusion set equipped with a 0.2μm or 0.22μm in-line filter must be used for administration.

      -The same infusion set must not be used for simultaneous administration of other drugs.

      -The diluted product should be administered immediately. If immediate use is not possible, the solution may be stored at room temperature for up to 4 hours (including storage in the infusion bag and infusion duration) or under refrigeration (2-8°C) for up to 24 hours (starting from the time of dilution). If refrigerated, allow the solution to reach room temperature prior to administration. Freezing the product is strictly prohibited.
   5. Prevention and Management of Infusion Reactions Previous studies indicate that infusion reactions may occur with drugs similar to IMM01. These reactions are associated with factors such as the subject's body type, age, concomitant diseases, aseptic techniques during infusion, and infusion rate. Infusion reactions, particularly allergic reactions, can progress rapidly and pose life-threatening risks, necessitating close attention.

      During infusion, investigators must closely monitor the patient's vital signs and observe for symptoms such as injection site reactions, rash, dizziness, headache, arthralgia, gastrointestinal disturbances, subcutaneous bleeding, itching, palpitations, chest tightness, nausea, vomiting, black stools, hematuria, and changes in mental status.

      Any patient discomfort must be addressed immediately, and detailed records should be maintained.

      If mild to moderate allergic reactions (e.g., urticaria, itching, fever, chills) occur during infusion, administration must be suspended immediately. The investigator will determine whether to resume infusion after the patient recovers, potentially reducing the infusion rate and extending the infusion duration as deemed appropriate. If no pre-infusion prophylactic medications were administered, glucocorticosteroids, antihistamines, antipyretics, or analgesics may be administered under close observation.
   6. Preventive Measures and Emergency Treatment Plan for Anaphylaxis of Trial Drugs Anaphylaxis, a severe and potentially life-threatening allergic reaction, represents a critical emergency in clinical immunology. It is characterized by a sudden onset of severe clinical symptoms involving multiple organ systems, mediated by immune or non-immune mechanisms, and triggered by various factors with diverse pathogenic pathways. Pathological features of fatal anaphylaxis include acute pulmonary hyperinflation, laryngeal edema, intra-alveolar hemorrhage, visceral congestion, pulmonary edema, and urticaria. Since all protein-based products carry the risk of inducing anaphylaxis, it is essential to establish an emergency treatment plan prior to initiating clinical trials. Research physicians and nurses must be thoroughly trained in the treatment protocol, proficient in all aspects of management, and regularly assessed by the research center to ensure prompt and appropriate intervention in the event of anaphylaxis.

In this study, detailed preventive measures and emergency treatment plans for allergic reactions to the investigational drug were established as follows:

1. The first and second doses for each subject should ideally be administered in the rescue room. The study physician must notify the anesthesiologist one day prior to administration.
2. Prior to drug administration, the research nurse must prepare emergency medications and equipment, reconfirm the subject's history of food or drug allergies, and educate the subject on potential infusion-related reactions. These may include injection-site reactions (e.g., redness, burning, swelling, pain), systemic symptoms (e.g., fever, chills, headache, itchy skin, rashes, throat itching, coughing, tachycardia, palpitations, chest tightness, dyspnea, dizziness, arthralgia, gastrointestinal disturbances), and changes in mental status. This ensures subjects remain vigilant and facilitates close monitoring during infusion.
3. If cardiac monitoring equipment is not used, measure vital signs every 15 minutes during the first 2 hours before the initial infusion, and at 2, 3, and 4 hours thereafter.
4. During infusion, the study nurse must remain with the subject, and the study physician should conduct assessments every 15-30 minutes.
5. If signs of an infusion reaction occur, immediately discontinue the infusion, measure blood pressure, notify the physician, and closely monitor the subject's condition.
6. The research physician must promptly assess the subject's condition based on clinical manifestations and initiate appropriate treatment. For complex or critical cases, the department head must be notified simultaneously. In the event of an acute allergic reaction, place the subject in a prone or head-down position, ensure airway patency and oxygenation, establish at least two intravenous lines for rapid fluid resuscitation, and administer anti-allergic medications (e.g., hydrocortisone sodium succinate, dexamethasone, 10% calcium gluconate, epinephrine, ipecac) as directed. Immediately notify the anesthesiologist to prepare for endotracheal intubation.
7. Continuously monitor the subject's condition until vital signs stabilize.
8. Provide reassurance to the subject and their family members.
9. Upon completion of resuscitation, the physician must promptly document the resuscitation details.

   7) Specific Immune-Mediated Adverse Reactions Immune-mediated adverse reactions, including severe and fatal cases, have been reported in patients treated with adebrelimab. These reactions may occur during or after discontinuation of therapy and can affect any organ system.

   Suspected immune-mediated adverse reactions must be evaluated and managed by a physician to exclude alternative etiologies. Most immune-mediated adverse reactions are reversible and can be managed by temporarily discontinuing the drug, initiating corticosteroid therapy, and/or providing supportive care. Therapy should be withheld for most Grade 2 and select Grade 3 and 4 immune-mediated adverse reactions. Permanent discontinuation is required for Grade 4 and select Grade 3 immune-mediated adverse reactions. For Grade 3 and 4 and select Grade 2 immune-mediated adverse reactions, administer 1-2 mg/kg/day prednisone (or equivalent) and other therapies as clinically indicated until symptoms improve to ≤ Grade 1.

   Corticosteroids should be tapered gradually over at least one month to prevent worsening or recurrence of adverse reactions. If symptoms persist or worsen despite corticosteroid therapy, non-corticosteroid immunosuppressive therapy should be initiated.

   Permanent discontinuation is required if any of the following occur: recurrent Grade 3 immune-mediated adverse reactions, failure to improve Grade 2 or 3 immune-mediated adverse reactions to Grade 0-1 within 12 weeks of the last dose (excluding endocrine disorders), or inability to taper corticosteroids to ≤10 mg/day prednisone equivalents within 12 weeks of the last dose.

   In cases of cytokine release syndrome (CRS), refer to the 2020 CSCO Guidelines for the Management of Malignant Hematologic Diseases.

   4. Treatment and Follow-Up No concomitant treatments are permitted in this study except for trametinib and Adebrelimab interventions. However, investigators must provide appropriate management based on the subject's clinical condition.

   Assessments will be conducted monthly for the first three months of treatment, followed by every three months thereafter. Additional assessments will occur at 3 months, 6 months, 1 year, 2 years, and 3 years after drug discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis and Grouping Criteria for LCH: Pathological confirmation of LCH via lesion biopsy, with positive immunohistochemistry for CD1a and/or CD207 (Langerin). Diagnostic and grouping criteria adhere to the 2009 standards established by the International Organization Cell Association and the CCHG-LCH-2019 research protocol by the Chinese Children's Histiocyte Group (CCHG). Disease assessment and treatment efficacy are evaluated based on the criteria set by the Society of Tissue and Cell Biology and the CCHG-LCH-2019 protocol. Treatment efficacy is categorized as: (1) No Active Disease (NAD); (2) Active Disease Better (AD-B); (3) Active Disease Stable (AD-S); (4) Active Disease Intermedia (AD-I); (5) Active Disease Worse (AD-W); (6) Relapse: Recurrence of new lesions after achieving NAD, AD-B, or AD-S, following maintenance treatment for over 3 months; (7) Refractory Disease: For SS-LCH patients, if the evaluation after first-line treatment results in AD-I or AD-W, and second-line treatment with cladribine or clofarabine still yields AD-I or AD-W; or MS-LCH patients with AD-I or AD-W after first-line treatment.

   Treatment responses are classified into three categories: favorable response (NAD and AD-B), moderate response (AD-I and AD-S), and adverse response (disease progression or relapse). The overall response rate (ORR) is defined as the percentage of patients achieving a favorable response (NAD or AD-B) at the evaluation time point among all enrolled patients.
2. Refractory or Recurrent LCH Criteria: Cases must meet at least one of the criteria for refractory or recurrent LCH.
3. Age Criteria: Initially, patients aged 6-17 years were included; subsequently, the age range was expanded to 1-17 years.
4. Informed Consent: All patients or their legal guardians must provide signed informed consent.
5. Performance Status: ECOG Performance Status (PS) score of 0-1; alternatively, a Karnofsky/Lansky Performance Status Scale score ≥ 50%.
6. Expected Survival: Minimum expected survival time of ≥ 6 months.
7. Organ Function Requirements:

   1. Cardiac Function: Left ventricular ejection fraction ≥ 50% on echocardiography, with no significant abnormalities on electrocardiogram.
   2. Renal Function: Serum creatinine ≤ 2.0 × ULN.
   3. Hepatic Function: ALT and AST ≤ 5.0 × ULN; total bilirubin ≤ 2.5 × ULN (≤ 3.0 × ULN for Gilbert syndrome). For patients with histiocytosis-related liver disease, abnormal bilirubin, AST, ALT, and albumin levels are permissible.
   4. Bone Marrow Function: Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L, hemoglobin ≥ 80 g/L (red blood cell transfusion allowed), and platelets ≥ 75 × 10^9/L (transfusion-independent, defined as no platelet transfusion within 7 days prior to enrollment).
   5. Oxygenation Status: Blood oxygen saturation > 91% in room air.

Exclusion Criteria:

1. Prior use of monoclonal antibodies or targeted therapies similar to anti-PD-1 or anti-PD-L1 agents.
2. Concurrent participation in other clinical trials.
3. Persistent treatment-related toxicity > Grade 1 (per CTCAE V5.0 criteria), excluding alopecia and neurotoxicity.
4. Known hypersensitivity to the active ingredients or excipients of trametinib and/or Adebrelimab.
5. History of autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, or Hashimoto's thyroiditis.
6. History of or current active tuberculosis infection.
7. Active infections requiring systemic treatment.
8. Severe comorbid conditions, including but not limited to uncontrolled diabetes or active peptic ulcer disease.
9. Positive serology for HIV, TP, HCV antibodies, HBV Ag, or HBV DNA copy number exceeding the upper limit of normal.
10. Thyroid dysfunction (abnormal FT3, FT4, T3, or T4 levels).
11. Administration of live or attenuated vaccines within 4 weeks prior to treatment initiation, during treatment, or within 5 months after the last dose.
12. Any condition deemed by the investigator to render the patient unsuitable for the study.
13. Inability or unwillingness to comply with the study protocol due to personal reasons.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-08-06 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Score | Before the 1st, 2nd, 3rd, 4th, 5th, and 6th cycles(each treatment cycle consists of four weeks), 1 week after discontinuation, 3 months, 6 months, 1 year, 2 years, 3 years
  The Disease Activity Score included the following parameters: bone pain, compression of other organs (orbits or spine), fever >38.5°C, lung imaging findings (pneumothorax, interstitial lesions), lung function (mechanical ventilation, pulmonary function tests [PFTs], oxygenation status, cyanosis), percentage of skin area affected, maximum diameter of soft tissue tumors (cm), presence of nodules >2 cm, liver location (below or above the umbilicus or no enlargement), spleen enlargement (assessed using the same criteria as the liver), hepatic enzymes >10 times the upper limit of normal, gamma-glutamyl transpeptidase (GGT) >10 times the upper limit of normal, serum albumin (g/L), platelet count, and hemoglobin (g/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided